CLINICAL TRIAL: NCT03064503
Title: Myocardial Fibrosis and Changes of Myocardial Function Related to Aging
Brief Title: Myocardial Fibrosis, Function and Aging
Acronym: MARVEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0744
Record Dates: First submitted 2017-02-21; First posted 2017-02-27 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: myocardial fibrosis; cardiac function; ageing
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): Sedentary healthy subjects will be recruited in this study. MRI, skin auto-fluorescence measures and blood sampling will be performed
  Interventions: Biological: Blood sampling; Device: MRI; Biological: Skin auto-fluorescence

INTERVENTIONS:
Biological: Blood sampling — Blood sampling will be performed at inclusion to investigate some biological eligibility criteria, and the day of MRI in order to analyse fibrosis biomarkers and collagen synthesis biomarkers
Device: MRI — MRI will be performed to measure interstitial fibrosis
Biological: Skin auto-fluorescence — Skin auto-fluorescence measures will be performed to measure advanced glycation end-products (AGE) produced by collagen degradation

SUMMARY:
In normal ageing, the impact of myocardial fibrosis on myocardial function is unclear as diastolic function is reported to change according to age. The objective is to explore the relationship between myocardial function changes, with local (T1 and diffusion) fibrosis measures with Magnetic Resonance Imaging (MRI) as well as global measures of fibrosis (skin auto-fluorescence and collagen blood-biomarkers).

ELIGIBILITY:
Inclusion Criteria:

* physical activity ≤ 3 x(30') per week
* no history of smoking, diabetes, myocardial infarction, heart failure, hypertension (<140 or <90 mmHg) and no anti-hypertensive or cardiovascular-related medications
* no familial history of early myocardial ischemia
* body mass index (BMI) <30kg/m2
* normal routine lipid blood analysis
* glycemia <1.26g/l
* normal electrocardiogram (ECG)

Exclusion Criteria:

* arrhythmia
* hepatic insufficiency
* pregnancy
* claustrophobia
* MRI contrast allergy,
* general contraindications to MRI such as pacemaker, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Regional myocardial strain | The day of MRI
  Segmental measures of systolic and diastolic strains with magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
MRI T1 value | The day of MRI, before gadolinium injection
  This value is an indicator of interstitial fibrosis and extracellular volume
MRI T1 value | The day of MRI, 15 minutes after gadolinium injection
  Diminution of this value after gadolinium injection is an indicator of increasing quantity of interstitial fibrosis and extracellular volume
Apparent Diffusion Coefficient (ADC) with MRI | The day of MRI
  ADC is measured with diffusion weighted imaging
Blood carboxy-terminal propeptide of procollagen type I (PICP) rate | The day of MRI
  Collagen blood biomarker analysis
Blood amino-terminal propeptide of procollagen type III (PIIINP) rate | The day of MRI
  Collagen blood biomarker analysis
Advanced Glycation End-products (AGE) rate | The day of MRI
  Skin auto-fluorescence AGE measures

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CROISILLE, MD, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Département de Radiologie, CHU Saint-Etienne - Hôpital Nord, Saint-Etienne, France